CLINICAL TRIAL: NCT01914003
Title: A Multi-Center Study of the Prevalence of Known Congenital Sucrase-Isomaltase Deficiency (CSID) Genetic Variants and Functional Sucrase Activity by 13C-Sucrose Breath Test in Children With Chronic Diarrhea or Chronic Abdominal Pain
Brief Title: Congenital Sucrase-Isomaltase Deficiency (CSID) Genetic Prevalence Study (GPS)
Acronym: CSID GPS
Status: Completed | Type: Observational
Sponsor: QOL Medical, LLC (Industry)
Collaborators: Arnold Palmer Hospital for Children (Other); Baylor College of Medicine (Other); Nationwide Children's Hospital (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); University of Mississippi Medical Center (Other); Children's Hospital and Research Center at Oakland (Unknown); Columbia University (Other); Children's Hospital Los Angeles (Other); Children's Hospital and Health System Foundation, Wisconsin (Other); Children's Center for Digestive Healthcare, LLC (Unknown); Massachusetts General Hospital (Other); Duke University (Other); Johns Hopkins University (Other); Children's Hospital of Philadelphia (Other); Children's Mercy Hospital Kansas City (Other); Children's Hospital Colorado (Other); Riley Children's Hospital (Unknown); Primary Children's Hospital (Other); State University of New York - Downstate Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: S2002
Record Dates: First submitted 2013-07-22; First posted 2013-08-01 (Estimated); Results first posted 2016-10-10 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2016-08

CONDITIONS: Congenital Sucrase-isomaltase Deficiency (CSID)
MeSH Terms: conditions — Sucrase-isomaltase deficiency, congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CSID Mutations: Individual has one or more known CSID mutations.
- Control: Individual does not have any known CSID mutations.

SUMMARY:
Congenital sucrose-isomaltase deficiency (CSID) is a rare, genetic disease in which mutations in the sucrose-isomaltase (SI) gene cause digestion problems of sucrose resulting in diarrhea and abdominal pain. Children with chronic, idiopathic diarrhea or abdominal pain will have their sucrose-isomaltase gene assessed for a panel of known CSID mutations to determine the prevalence of these mutations in an enriched population and also determine functional deficiency using a breath test.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or younger.
* A primary clinical diagnosis of chronic idiopathic diarrhea or chronic abdominal pain for at least 4 weeks.
* English or Spanish speaking subjects and parent(s)/guardian only.
* Parental consent from one parent/guardian and also subject assent when appropriate based on individual IRB requirements.

Exclusion Criteria:

* Any condition(s) or finding(s) that in the opinion of the principal investigator suggests an alternative diagnosis for his/her gastrointestinal symptoms.
* Abdominal pain primarily related to constipation.
* Suspected gastrointestinal infectious disease.
* No current use of sacrosidase (Sucraid® Oral Solution).
* Known gastrointestinal disease such as celiac disease.
* Prior consumption of an investigational medication within the last 4 weeks.
* Antibiotics in the last 2 weeks, and no history of viral gastroenteritis within that same period of time.
* Known Hepatitis B or C infection (positive HBsAg or HCV within 6 months of enrollment) or Subject-Pugh Class C liver disease of any cause, HIV infection, tuberculosis, Clostridia difficile co-infection, cancer or systemic infections.
* Severe neurologic impairment that would prevent them from reporting a history of abdominal pain.
* Receiving or received biologic therapies (including infliximab, adalimumab, natalizumab) within 3 months prior to or at enrollment.
* Present or past use of immune modulators therapy (e.g., azathioprine, 6MP, methotrexate).
* Planned or previous abdominal surgery (e.g., bowel resection).
* Subjects with severe, uncontrolled systemic diseases.
* Presence of clinical alarm signs, including hypotension, anemia requiring blood transfusions, altered mental status, or inability to tolerate food and/or fluids by mouth.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 18 years of age or younger experiencing chronic, idiopathic diarrhea or abdominal pain for at least 4 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2013-05; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital and Research Center of Oakland, Oakland, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - Arnold Palmer Children's Hospital, Orlando, Florida
  - Children's Center for Digestive Healthcare, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Johns Hopkins Children's Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Morgan Stanley Children's Hospital, New York, New York
  - Stony Brook University, Stony Brook, New York
  - Duke University Children's Hospital, Durham, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- See also: Study overview — http://www.csidgps.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CSID Mutations | Control
Started | 27 | 26
Completed | 19 (Number of subjects who completed through study and qualify as evaluable) | 14 (Number of subjects who completed through study and qualify as evaluable)
Not Completed | 8 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CSID Mutations | Control | Total
Number analyzed (Participants) | 27 | 26 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 27 | 26 | 53
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 8 [1 to 13] | 10.5 [6.25 to 16] | 9 [2 to 15]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 13 | 10 | 23
Region of Enrollment [Number; unit: participants]
  United States | 27 | 26 | 53

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of CSID Genetic Variants
Description: Prevalence of CSID genetic variants in subjects 18 years of age or younger with a primary symptom of chronic idiopathic diarrhea or chronic abdominal pain without constipation.
Time Frame: 1 year
Measure: Number; unit: Participants
Arm/Group | CSID Mutations | Control
Number analyzed (Participants) | 27 | 26
Participants | 27 | 0

ADVERSE EVENTS:
Time Frame: Monitoring for adverse events occurred throughout the study, but none were expected or reported as no study drug was involved and minimally invasive procedures were used to obtain genetic and breath samples.
Arm/Group | CSID Mutations | Control
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/26
Other Adverse Events (participants affected / at risk) | 0/27 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
As outlined in each Clinical Trial Agreement between Sponsor and PI.